CLINICAL TRIAL: NCT05798234
Title: Factors Associated With Failure of HFNO in COVID-19 ICU Patients
Acronym: CO-OHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI120
Record Dates: First submitted 2023-04-03; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: high flow oxygen device — no intervention

SUMMARY:
To determine the factors associated with OHD failure in COVID-19 patients admitted to an Intensive Care Unit

DETAILED DESCRIPTION:
Patients admitted into 1 participating ICU for acute hypoxemic respiratory failure due to COVID-19 between 02/01/2020 and 06/01/2022 will be assessed for OHD failure

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in ICU for COVID-19 pneumonia

Exclusion Criteria:

* under immediate ECMO
* secondary transferred from another ICU
* readmission in the ICU
* initial limitation of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
High flow oxygen failure | icu stay duration
  patients requiring initial high flow oxygen but finally intubated

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Médicale, Hôpital Central, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided
undecided